CLINICAL TRIAL: NCT02157012
Title: Evaluation of the Condition After Xeljanz Treatment in Rheumatoid Arthritis Patients
Brief Title: Evaluation of the Condition of Rheumatoid Arthritis After Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shinshu University (Other)
Collaborators: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Assistant Professor, Shinshu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Xeljanz2014
Record Dates: First submitted 2014-06-01; First posted 2014-06-05 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- The condition of rheumatoid arthritis (Experimental)
  Interventions: Drug: The effectiveness of Xeljanz in rheumatoid arthritis patients

INTERVENTIONS:
Drug: The effectiveness of Xeljanz in rheumatoid arthritis patients

SUMMARY:
To examine the safety and effectiveness after Xeljanz treatment in rheumatoid arthritis patients

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis

Exclusion Criteria:

* Other connective tissue disease

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of clinical evaluation in rheumatoid arthritis | Every month
  DAS28, SDAI, Blood testing, Plain radiograph, and Ultrasound will be performed.

SECONDARY OUTCOMES:
Number of participants with adverse events | Every month

CONTACTS AND LOCATIONS:
Locations (1):
- Yukio Nakamura, Matsumoto, Nagano, Japan